CLINICAL TRIAL: NCT01543828
Title: A Phase IV, Randomized, Double-blind, Placebo-controlled, Multicenter, Exploratory, Single-dose Crossover Study With Indacaterol 75 μg Compared to Placebo, Assessing Time to Patient's Perception of Onset of Effect in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: Indacaterol 75 μg Compared to Placebo, Assessing Time to Patient's Perception of Onset of Effect in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149BUS01
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: COPD
Keywords: COPD; Indacatarol; placebo; crossover; patient perception
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- indacaterol then placebo (Experimental): In treatment 1: participants received indacaterol 75 µg one dose delivered via single-dose dry-powder inhaler (SDDPI) followed by treatment 2: placebo one dose via SDDPI between day 7 and 10. Albuterol was available for use as rescue medication.
  Interventions: Drug: indacaterol
- placebo then indacaterol (Placebo Comparator): In treatment 1, participants received placebo one dose delivered via SDDPI followed by treatment 2: indacaterol 75 µg one dose delivered via SDDPI between Day 7 and Day 10. Albuterol was available for use as rescue medication.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: indacaterol — delivered via single-dose dry-powder inhaler
  Arms: indacaterol then placebo
Drug: placebo — delivered via single-dose dry-powder inhaler
  Arms: placebo then indacaterol

SUMMARY:
This is a phase IV study of indacaterol 75 μg single-dose compared to placebo in moderate-severe COPD patients with breathing symptoms to assess time to patient's perception of onset of effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a COPD exacerbation requiring systemic corticosteroids and/or antibiotics and/or hospitalization in the 6 weeks prior to screening
* Diagnosis of chronic obstructive pulmonary disease (COPD) (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease [GOLD] Guidelines, 2008) and:

  * Smoking history of at least 10 pack-years
  * Post-bronchodilator forced expiratory volume in 1 second (FEV1) ≤ 70% and ≥ 40% of the predicted normal value
  * Post-bronchodilator FEV1/FVC (forced vital capacity) < 70%
  * Breathing symptoms that interfere with daily activities

Exclusion Criteria:

* Patients who have had a COPD exacerbation requiring systemic corticosteroids and/or antibiotics and/or hospitalization in the 6 weeks prior to screening
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients who require oxygen therapy for chronic hypoxemia, are receiving bronchodilators or other medications for COPD that are dosed once daily, are unable to follow instruction on rescue albuterol use during the study, or are at risk deterioration of COPD with study procedures. Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with uncontrolled diabetes mellitus
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular co-morbid conditions

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (6):
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Period: Treatment 1
Arm/Group | Indacaterol Then Placebo | Placebo Then Indacaterol
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Treatment 2
Arm/Group | Indacaterol Then Placebo | Placebo Then Indacaterol
Started | 20 | 19 (1 participant completed treatment 1, had an adverse event, and did not receive treatment 2.)
Completed | 19 | 19
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol Then Placebo | Placebo Then Indacaterol | Total
Number analyzed (Participants) | 20 | 20 | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 62.2 (10.29) | 60.8 (6.90) | 61.5 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 11 | 16 | 27

OUTCOME MEASURES:

1. Primary Outcome: Time (in Minutes) to Patient's Perception of Onset of Effect
Description: Defined as the first time point that the patient responds "yes" to the following self-administered question:
  "I feel that the drug is working in improving my breathing?"
Time Frame: 5, 7.5, 10, 15, 20, 30, 40, 50, and 60 minutes post dose for treatment 1 and treatment 2
Population: Full Analysis Set included all participants who received one dose of study drug.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- indacaterol_treatment 1: In treatment 1: participants received indacaterol 75 µg one dose delivered via single-dose dry-powder inhaler (SDDPI). Albuterol was available for use as rescue medication.
- indacaterol_treatment 2: In treatment 1, participants received placebo one dose delivered via SDDPI followed by treatment 2: indacaterol 75 µg one dose delivered via SDDPI between Day 7 and Day 10. Albuterol was available for use as rescue medication.
- placebo_treatment 1: In treatment 1, participants received placebo one dose delivered via SDDPI. Albuterol was available for use as rescue medication.
- placebo_treatment 2: In treatment 1: participants received indacaterol 75 µg one dose delivered via single-dose dry-powder inhaler (SDDPI) followed by treatment 2: placebo one dose via SDDPI between day 7 and 10. Albuterol was available for use as rescue medication.
Arm/Group | indacaterol_treatment 1 | indacaterol_treatment 2 | placebo_treatment 1 | placebo_treatment 2
Number analyzed (Participants) | 20 | 19 | 20 | 20
Minutes | 25.13 (27.726) | 26.05 (28.787) | 21.88 (25.928) | 25.88 (27.449)

ADVERSE EVENTS:
Groups:
- Indacaterol: Participants received indacaterol 75 µg one dose delivered via single-dose dry-powder inhaler (SDDPI).
- Placebo: Participants received placebo one dose delivered via SDDPI.
Arm/Group | Indacaterol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 2/40 | 0/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol (N=40) | Placebo (N=40)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.